CLINICAL TRIAL: NCT01971840
Title: Effectiveness of an Intervention of Physical Activity Promotion in Schoolchildren on Preventing Obesity During the Adiposity Rebound Period: a Cross-over Randomized Cluster Trial.
Brief Title: Effectiveness of a Physical Activity Intervention on Preventing Obesity During the Adiposity Rebound Period.
Acronym: MOVI-KIDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, FRANCISCO QUILES VICECHANCELLOR OF RESEARCH, Proffesor / PhD, University of Castilla-La Mancha
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PI12/02400
Record Dates: First submitted 2013-10-07; First posted 2013-10-29 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-10

CONDITIONS: Physical Activity; Adiposity; Children; Obesity; Cardiovascular Disease
Keywords: Physical activity; Physical fitness; Obesity; Adiposity; Adiposity rebound period; Children; Blood pressure; Randomized controlled trials; Barriers and facilitators of the environment
MeSH Terms: conditions — Motor Activity; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MOVI-KIDS Program (Experimental): Intervention group
  Interventions: Behavioral: MOVI-KIDS
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: MOVI-KIDS — MOVI-KIDS is a multidimensional intervention that consist of: a) for children, 4.5 h/week of a standardized recreative, non-competitive physical activity extracurricular program; b) informative sessions to parents and teachers about how schoolchildren can became more active, and c) interventions in the playground (environmental changes: equipment, facilities, painting, etc.) aimed to promote physical activity during recess (MOVI-Playground).
  Arms: MOVI-KIDS Program

SUMMARY:
Coordinated project whose objectives are: a) to assess the effectiveness of a physical activity intervention (MOVI-KIDS) on preventing obesity and improving fitness during the adiposity rebound period; and b) to examine the effectiveness of MOVI-KIDS on reducing the carotid intima-media thickness.

DETAILED DESCRIPTION:
The prevalence of overweight in Spanish children in the puberty age is among the highest in the world and increasing quickly. Our group has done so far two interventions based on after-school programs of recreational physical activity to control obesity and other cardiovascular risk factors in primary school children (8-to-11 years)in Cuenca, Spain.

The first edition, called MOVI, showed moderate effect in reducing adiposity and improving the lipid profile, but did not significantly improve overall cardiometabolic risk, mainly because of did not reduce blood insulin levels. A second edition (MOVI-2), increased duration and intensity of the sessions and was more focused on increased muscle strength. Preliminary analysis also show a decrease in body fat, a reduction of global cardiometabolic because of decreased insulin levels.

Our project integrates a multidimensional intervention to promote physical activity, with a mixed design (cross-over randomized trial, and a qualitative study) and consist of two sub-projects that share the same study population: "Effectiveness of an intervention of physical activity promotion in schoolchildren on preventing obesity during the adiposity rebound period: a cross-over randomized cluster trial" and "Effectiveness of physical activity intervention to prevent obesity and improve academic performance in children with and without ADHD risk".

The two interventions are based on a cross-over randomized trial aimed to test the effectiveness of an intervention to promote physical activity in the school environment (MOVI-KIDS) during two-years in 22 schools (20 public and two private schools) in the provinces of Cuenca and Ciudad Real, Spain.

This principal subproject consisted of a mixed study including both the trial cited above and a nested qualitative study aimed to identify barriers and facilitators to physical activity in children in the school environment (social and family factors, urban planning, etc.), and produce knowledge about the perceptions of children, parents and teachers on how you can improve conditions of physical and social environment to facilitate physical activity.

The hypotheses of this third edition are that a multidimensional intervention promoting physical activity in children at the adiposity rebound period (4-7 years),in the school environment (MOVI-KIDS), lasting two-years, will to:

1. Reduce the body fat percentage in the intervention group versus the control group in 2%.
2. Improve the several components of fitness: aerobic capacity, strength, speed and agility.
3. Reduce the carotid intima-media thickness and
4. Reduce fat, increase fat free mass, and reduce sedentary behavior.

ELIGIBILITY:
Inclusion Criteria:

* Schools with at least one full course of 3rd of early childhood education and one of 1st primary school.
* The Boards of Governors (community participatory organ in each school) give its approval to the intervention and measurements at the beginning and end of the course.
* Children 4 to 7 years old.
* Children's parents/caregivers will give their written consent to the children's participation.
* Collaboration in the family to respond to questionnaires on family leisure habits, sleeping, eating, getting around town, etc., included in the measurement protocol of this project.

Exclusion Criteria:

* Have a malformation that prevents learning of the Spanish language (or Spanish sign language).
* Have some kind of physical or mental disorder identified by parents or teachers that prevent physical activity.
* Have a chronic illness such as heart disease, diabetes or asthma, as determined by your pediatrician/family doctor -after analysis of the activities program- prevents participation in them.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1600 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Body fat percentage | One year (interim analysis)
  To reduce body fat percentage in the intervention group versus the control group in 2% in children during the adiposity rebound 4-7 years).
  Mean of two measurements of body fat percentage using an eight-electrode BC-418 MA bioimpedance analysis system (Tanita Corp. Tokyo, Japan).

SECONDARY OUTCOMES:
Physical fitness | One year (interim analysis)
  It will be assessed the main components of fitness: a) muscle strength by using standing long jump test b) Flexibility by using the sit and reach test c) speed-agility (The 4x10 meters shuttle run test), d) aerobic capacity, by using 20-m shuttle run test, which is validated to measure maximal aerobic capacity in children from 5 years.
Waist circumference | One year (interim analysis)
  Waist circumference will be measured 3 times at the midpoint between the last rib and the iliac crest at the end of a normal expiration and using a flexible tape.
Tricipital skinfold thickness | one year (interim analysis)
  Skinfold thickness will be measured 3 times at the triceps using a Holtain Ltd. caliper (0.2 mm accuracy and consistent 10 g/mm2 pressure between valves)
Blood pressure | one year (interim analysis)
  Blood pressure will be measured twice, with a 5-min interval between measurements. The first measurement will be made after at least 5 min rest. The child will be seated, in relaxing conditions, with the right arm semi-flexed at heart level. Blood pressure will be measured with an Omron M5-I monitor (Omron Healthcare UK Ltd.) using one of 3 different cuff sizes according to arm circumference.

OTHER OUTCOMES:
Prior assessment of barriers and facilitators | One year
  Nested qualitative study aimed to understand the barriers and limitations perceived by children, parents, and teachers for the physical activity of schoolchildren, using focus groups under a phenomenologic framework.

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Martínez-Vizcaíno, PhD, Principal Investigator — Health and Social Research Centre, University of Castilla-La Mancha, Cuenca, Spain
Locations (1):
- Health and Social Research Centre, University of Castilla-La Mancha, Cuenca, Cuenca, Spain

REFERENCES:
- [Derived] Martinez-Vizcaino V, Pozuelo-Carrascosa DP, Garcia-Prieto JC, Cavero-Redondo I, Solera-Martinez M, Garrido-Miguel M, Diez-Fernandez A, Ruiz-Hermosa A, Sanchez-Lopez M. Effectiveness of a school-based physical activity intervention on adiposity, fitness and blood pressure: MOVI-KIDS study. Br J Sports Med. 2020 Mar;54(5):279-285. doi: 10.1136/bjsports-2018-099655. Epub 2019 Jan 9. PMID 30626597
- [Derived] Pozuelo-Carrascosa DP, Sanchez-Lopez M, Cavero-Redondo I, Torres-Costoso A, Bermejo-Cantarero A, Martinez-Vizcaino V. Obesity as a Mediator between Cardiorespiratory Fitness and Blood Pressure in Preschoolers. J Pediatr. 2017 Mar;182:114-119.e2. doi: 10.1016/j.jpeds.2016.11.005. Epub 2016 Nov 29. PMID 27912924
- [Derived] Martinez-Vizcaino V, Mota J, Solera-Martinez M, Notario-Pacheco B, Arias-Palencia N, Garcia-Prieto JC, Gonzalez-Garcia A, Alvarez-Bueno C, Sanchez-Lopez M; MOVI-KIDS group. Rationale and methods of a randomised cross-over cluster trial to assess the effectiveness of MOVI-KIDS on preventing obesity in pre-schoolers. BMC Public Health. 2015 Feb 22;15:176. doi: 10.1186/s12889-015-1512-0. PMID 25884885
- See also: Information and results of the first and second edition of the MOVI Program — http://www.movidavida.org